CLINICAL TRIAL: NCT07087275
Title: Long-term Visual and Refractive Outcomes After Traumatic Cataract Surgery in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Jin Yang (Other)
Collaborators: The Eye Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor-Investigator, Jin Yang, Chief Physician, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Other Study IDs: Traumatic Cataract-FDU-2010
Record Dates: First submitted 2025-07-05; First posted 2025-07-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Cataract
Keywords: Traumatic Cataract; Cataract Surgery; Pediatric Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic cataract: Traumatic cataract

SUMMARY:
This prospective multicenter observational study aims to evaluate long-term visual and ocular biometric outcomes in pediatric patients aged 0-16 years who were diagnosed with traumatic cataract and underwent cataract extraction surgery. Medical records of eligible patients with at least 5 to 10 years of postoperative follow-up will be reviewed. Key outcome measures include best-corrected visual acuity (BCVA), axial length, corneal astigmatism, intraocular pressure (IOP), binocular function (fusion and stereopsis), intraocular lens (IOL) position, and postoperative complications. The study seeks to provide insight into long-term visual rehabilitation and prognostic indicators following pediatric traumatic cataract surgery.

ELIGIBILITY:
Inclusion Criteria

1. Aged 0 to 16 years at the time of trauma-related cataract diagnosis
2. Diagnosed with traumatic cataract (due to blunt or penetrating ocular trauma)
3. Underwent cataract extraction surgery with or without intraocular lens (IOL) implantation
4. Able to attend regular follow-up assessments for at least 5 years postoperatively
5. Written informed consent obtained from a parent or legal guardian

Exclusion Criteria

1. Congenital or developmental cataract
2. Pre-existing ocular diseases unrelated to trauma (e.g., congenital glaucoma, retinal dystrophies)
3. Severe posterior segment damage precluding reliable visual outcome evaluation (e.g., endophthalmitis, choroidal rupture involving the macula)
4. Systemic or neurological disorders that affect vision or compliance with follow-up (e.g., cerebral palsy, intellectual disability)
5. Previous intraocular surgery in the affected eye unrelated to the trauma

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will enroll pediatric patients aged 0 to 16 years who were diagnosed with traumatic cataract and underwent cataract surgery at the Eye, Ear, Nose, and Throat Hospital of Fudan University, or the Eye Hospital of Wenzhou Medical University, or the First Affiliated Hospital of Nanjing Medical University. Eligible patients may have experienced either blunt or penetrating ocular trauma. Both unilateral and bilateral cases are included. All participants must be able to complete regular follow-up evaluations for at least 5 years after surgery. The study population reflects a broad spectrum of post-traumatic cataract severity and treatment modalities, representing real-world clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | From surgery up to 10 years postoperatively, depending on available follow-up duration
  UDVA & BCVA will be assessed using age-appropriate optotypes (e.g., Lea symbols, Snellen chart, or ETDRS chart) and recorded in logMAR units.
Axial Length Development | From surgery up to 10 years postoperatively, depending on available follow-up duration
  Axial Length(mm) measured by IOLMaster700
Corneal Astigmatism | From surgery up to 10 years postoperatively, depending on available follow-up duration
  Measured by Pentacam
Corneal Astigmatism | From surgery up to 10 years postoperatively, depending on available follow-up duration
  Measured by IOLMaster700

SECONDARY OUTCOMES:
Binocular Function | From surgery up to 10 years postoperatively, depending on available follow-up duration
  Binocular fusion and stereopsis will be assessed using standard clinical tools such as Worth 4-dot test and Randot stereoacuity test.
Intraocular Pressure (IOP) | From surgery up to 10 years postoperatively, depending on available follow-up duration
  IOP(mmHg) will be monitored using non-contact or Goldmann applanation tonometry to detect postoperative ocular hypertension or glaucoma.
Postoperative Complications | From surgery up to 10 years postoperatively, depending on available follow-up duration
  Incidence of complications such as secondary glaucoma, visual axis opacification, retinal detachment, or IOL decentration will be recorded.
Intraocular Lens (IOL) Position | From surgery up to 10 years postoperatively, depending on available follow-up duration
  IOL centration and tilt will be evaluated by slit-lamp exam or anterior segment OCT.
Anterior Chamber Depth (ACD) | From surgery up to 10 years postoperatively, depending on available follow-up duration
  Anterior chamber depth (ACD) will be measured using optical biometry and recorded in millimeters (mm) as the distance from the corneal endothelium to the anterior lens surface.
Lens Thickness (LT) | From surgery up to 10 years postoperatively, depending on available follow-up duration
  Lens thickness (LT) will be measured using optical biometry and recorded in millimeters (mm).
White-to-White Corneal Diameter (WTW) | From surgery up to 10 years postoperatively, depending on available follow-up duration
  WTW corneal diameter will be measured using optical biometry and recorded in millimeters (mm).
Keratometry | From surgery up to 10 years postoperatively, depending on available follow-up duration
  Keratometric values will be measured using optical biometry and recorded in diopters (D).

CONTACTS AND LOCATIONS:
Locations (1):
- Eye and ENT hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No